CLINICAL TRIAL: NCT03600077
Title: Evaluation of Supra-aortic Trunks Debranching Techniques in Open Arch Repair by Means of Frozen Elephant Trunk Procedure With Two Configurations of the Jotec E-Vita Hybrid Graft
Brief Title: Evaluation of Supra-aortic Trunks Debranching Techniques in Open Arch Repair by Means of Frozen Elephant Trunk Procedure With Two Configurations of the Jotec E-Vita Hybrid Graft (FETOPT)
Acronym: FETOPT
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Bertoglio Luca, Principal Investigator, IRCCS San Raffaele
Other Study IDs: FETOPT/18/OSR
Record Dates: First submitted 2018-04-05; First posted 2018-07-26 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Aneurysms Aortic Arch
MeSH Terms: conditions — Aneurysm, Aortic Arch

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate two different supra-aortic trunks debranching techniques during open repair of aortic arch aneurysms by means of Frozen Elephant Trunk procedure with two configurations of the Jotec E-Vita hybrid graft.

DETAILED DESCRIPTION:
Open management of extensive pathology of the proximal aorta, namely ascending aorta, aortic arch, and descending thoracic aorta (DTA) requires sequential treatment of each segment involved. According to the etiopathogenesis and clinical history of the disease, each segment can be treated independently or in association with the other portions of diseased aorta.

The current standard of treatment for arch aneurysmal disease extending into the DTA is the elephant trunk technique: both conventional and "frozen". The first requires open repair of the aortic arch with the use of a conventional surgical graft which distal end is left dangling in the DTA and will be the site of the proximal anastomosis of the subsequent repair of the thoracic aneurysm. The frozen elephant trunk (FET) technique differs from the first for the graft employed: this graft has a distal stented portion which is deployed in the DTA and facilitates subsequent endovascular management of the thoracic pathology.

In both the conventional elephant trunk and frozen elephant trunk the supra-aortic trunks (innominate artery, left carotid artery and left subclavian artery) need to be reimplanted on the surgical graft with variable configurations.

Debranching and reimplantation of such vessels can occur with variable configurations and either before or after the substitution of the pathologic aorta which is performed during cardiac arrest and extra-corporeal circulation (ECC) The first design has a straight tubual graft with self-expanding stents in the distal portion and has been employed at department of Vascular Surgery in San Raffaele Hospital, from December 2009 to February 2016. The second design has two side-branches on the non-stented proximal portion which facilitate debranching of the supra-aortic trunks before cardiac arrest and allow early reperfusion of the visceral vessels during extra-corporeal circulation . This graft has been introduced in practice at department of Vascular Surgery at San Raffaele Hospital in November 2016.

The investigators review a prospectively compiled Microsoft Office Excel database with the procedural details of the 30 patients affected by extensive proximal aortic pathology treated at department of Vascular Surgery in San Raffaele Hospital between December 2009 and January 2017 by means of Frozen Elephant Trunk technique, and of those of the next 20 patients who will be treated with the same procedure.

ELIGIBILITY:
Inclusion Criteria:

patient undergoing treatment of extensive proximal aortic pathology at San Raffaele Hospital since December 2009

Exclusion Criteria:

extensive proximal aortic pathology treated by techniques other than frozen elephant trunk : total open aortic repair, total endovascular aortic repair, hybrid endovascular aortic repair in zone 0.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The Investigators review a prospectively compiled Microsoft Office Excel database with the procedural details of the 30 patients affected by extensive proximal aortic pathology treated at San Raffaele Hospital between December 2009 and January 2017 by means of Frozen Elephant Trunk technique, and of those of the next 20 patients who will be treated with the same procedure.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-07-19 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Extracorporeal circulation times (minutes) | Intraoperative
  - Extracorporeal circulation time
antegrade cerebral perfusion time (minutes) | Intraoperative
  - antegrade cerebral perfusion time
Lower limb perfusion time (minutes) | Intraoperative
  - Lower limb perfusion time

SECONDARY OUTCOMES:
Clinical 30-day results (Percent of participants with the clinical outcome) | Perioperative, 30 days
  - Mortality (%)
Clinical 30-day results (Percent of participants with the clinical outcome) | Perioperative, 30 days
  - Stroke (%)
Clinical 30-day results (Percent of participants with the clinical outcome) | Perioperative, 30 days
  - Spinal cord ischemia ( %)
Clinical 30-day results (Percent of participants with the clinical outcome) | Perioperative, 30 days
  - Prolonged mechanical ventilation: >48h ( %)
Clinical 30-day results (Percent of participants with the clinical outcome) | Perioperative, 30 days
  - Renal impairment (%)

CONTACTS AND LOCATIONS:
Locations (1):
- San Raffaele Hospital, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Di Eusanio M, Borger M, Petridis FD, Leontyev S, Pantaleo A, Moz M, Mohr F, Di Bartolomeo R. Conventional versus frozen elephant trunk surgery for extensive disease of the thoracic aorta. J Cardiovasc Med (Hagerstown). 2014 Nov;15(11):803-9. doi: 10.2459/JCM.0b013e328364559c. PMID 23867913
- [Result] Hagl C, Pichlmaier M, Khaladj N. Elephant trunks in aortic surgery: fresh and frozen. J Thorac Cardiovasc Surg. 2013 Mar;145(3 Suppl):S98-102. doi: 10.1016/j.jtcvs.2012.11.065. PMID 23410783
- [Derived] Bertoglio L, Fittipaldi A, Giambuzzi I, Redaelli P, Verzini A, Cambiaghi T, Bargagna M, Alfieri O, Chiesa R, Castiglioni A. Preliminary Results of Debranch-First Technique in Frozen Elephant Trunk Procedures. Ann Thorac Surg. 2019 Nov;108(5):1345-1353. doi: 10.1016/j.athoracsur.2019.04.010. Epub 2019 May 10. PMID 31082360